CLINICAL TRIAL: NCT06340802
Title: A First in hUman Study for Resistant Epilepsy With the Vagus Nerve stimulatiOn Device by syneRgia medicAl
Acronym: AURORA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synergia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SYG001
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Drug Resistant Epilepsy
Keywords: vagus nerve stimulation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VNS Treatment (Experimental): Vagus nerve stimulation is started 2-week after the implantation.
  Interventions: Device: VNS Treatment

INTERVENTIONS:
Device: VNS Treatment — Vagus nerve stimulation is started 2-week after the implantation

SUMMARY:
This is an open label, single arm, interventional, prospective first in human study, designed to evaluate the safety of the NAO.VNS SYSTEM.

DETAILED DESCRIPTION:
This is the first clinical investigation with the NAO.VNS SYSTEM from Synergia Medical.

Up to 10 patients with drug resistant epilespy, who are eligible for vagus nerve stimulation, will be included in two sites.

The total duration of the study is expected to be 36 months. Study procedures are composed of (i) baseline, (ii) implantation, (iii) titration and (iv) follow-up until 24 months.

Primary objective is to evaluate safety of the NAO.VNS SYSTEM.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the Informed Consent Form (ICF) and the study procedures and provide written consent or, in case of cognitive impairment, be the legal ward of a person who is able and willing to provide written consent.
2. Subjects diagnosed with Drug Resistant Epilepsy (DRE) and candidate for VNS treatment
3. Ability of subjects or, in the case of cognitive impairment, their caregiver, to accurately count seizures and complete seizure diaries.
4. Adult subjects, age ≥ 18.
5. Willingness of subjects or, in the case of cognitive impairment, their caregiver, to charge the NAO.VNS system with the Smart Charger on a weekly basis.
6. Subjects' willingness to follow the protocol procedures. For example, subject should have a careful seizure diary completion according to standard of care to ensure 8 weeks of data available by time of implant.
7. Female subjects of childbearing age using acceptable methods of birth control (abstinence considered acceptable).

Exclusion Criteria:

1. Unstable medical condition likely to precipitate seizures and make it difficult to evaluate efficacy.
2. Prior cervical vagotomy.
3. Progressive neurological disease.
4. Pregnancy.
5. Significant cardiac or pulmonary disease under treatment.
6. History of noncompliance for seizure diary completion.
7. Prior implant with vagus nerve stimulation device.
8. Current active treatment of epilepsy with cerebellar or thalamic stimulation.
9. Prior therapeutic brain surgery for epilepsy within the last 6 months prior to NAO.VNS implantation.
10. Receiving or likely to receive short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy after implantation.
11. Currently receiving another investigational treatment.
12. Patient with Vocal Cord Palsy (VCP), including unilateral, whatever the side.
13. Diabetic patients and all patients with a known vagal neuropathy.
14. Coagulation disorder, wound healing and bleeding disorder or taking anticoagulant medication (oral anticoagulants; antiplatelets (such as aspirin, ticagrelor) are allowed).
15. Patient currently participating in another clinical investigation, without explicit consent of the Sponsor (non-interventional registries are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | through 3 months of implantation
  Incidence rate of NAO.VNS device-related treatment emergent adverse events (TEAE)
Procedure and/or device related adverse events | through 30 days post implant
  Incidence of procedure and/or device related adverse events

SECONDARY OUTCOMES:
Device-related treatment emergent adverse events | through 6, 12, 18 & 24 months of implantation
  Incidence rate of NAO.VNS device-related treatment emergent adverse events
Device deficiencies | at 3, 6, 12, 18 and 24 months of implantation
  Number of physician reported device deficiencies related to NAO.VNS
Procedural Success | at implantation surgery
  Procedural Success defined as successful implantation of the device without the occurrence of procedure related serious adverse events (from incision to closure).
Change in seizure frequency | at 3, 6, 12, 18 & 24 months of implantation.
  Change in seizure frequency, as compared to preoperative baseline
Proportion of responders | at 3, 6, 12, 18 & 24 months of implantation
  Proportion of patients with at least a 50% reduction in the frequency of seizures, as compared to preoperative baseline
Change in seizure severity | at 3, 6, 12, 18 & 24 months of implantation
  Change in seizure severity, as compared to preoperative baseline, as measured by the "Seizure Severity Questionnaire" (SSQ)
Change in quality of life | at 3, 6, 12, 18 & 24 months of implantation
  Change in quality of life, as compared to preoperative baseline, as measured by the "QUALITY OF LIFE IN EPILEPSY" (QOLIE-31)
Changed in mood | at 3, 6, 12, 18 & 24 months of implantation
  Changed in mood, as compared to preoperative baseline, as measured by the "Beck Depression Inventory" (BDI)
Usability | at 3, 6, 12, 18 & 24 months of implantation
  Usability and workflow assessment evaluated through a practitioner's and patient's questionnaire

OTHER OUTCOMES:
Exploratory Endpoints | at 3, 6, 12, 18 & 24 months of implantation
  Number of successfull Laryngeal Muscle-Evoked Potential recordings during follow-up visits recorded by the NAO.VNS clinician programmer.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - Cliniques Universitaires St.-Luc, Brussels
  - UZ GENT (Universitair Ziekenhuis Gent), Ghent
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No